CLINICAL TRIAL: NCT03821415
Title: A Phase II, Multicentre, Randomised, Placebo-controlled, Doublemasked Trial of RP101 Ophthalmic Formulation Versus Vehicle in Post-menopausal Women With Moderate to Severe Dry Eye Syndrome
Brief Title: Effects of RP101 in Post-menopausal Women With Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Redwood Pharma AB (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP101-200
Record Dates: First submitted 2019-01-16; First posted 2019-01-29 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Dry Eye Syndromes
Keywords: Keratoconjunctivitis sicca; Dry Eye Disease; Slow-release; Ophthalmology; Topical Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised, double-masked, parallel-group, placebo-controlled Phase II study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 - RP101 0.05% (Experimental): RP101 0.05% (w/w) 17β-oestradiol-3-phosphate ophthalmic sterile solution, one drop each eye every 12 h (b.i.d.) for 90 consecutive days
  Interventions: Drug: RP101
- 2 - RP101 0.1% / Placebo (Experimental): RP101 0.1% (w/w) 17β-oestradiol-3-phosphate ophthalmic sterile solution, one drop each eye in the morning (q.d.) followed by one drop of placebo each eye in the evening for 90 consecutive days
  Interventions: Drug: RP101
- 3 - RP101 0.1% (Experimental): RP101 0.1% (w/w) 17β-oestradiol-3-phosphate ophthalmic sterile solution, one drop each eye every 12 h (b.i.d.) for 90 consecutive days
  Interventions: Drug: RP101
- 4 - Placebo (Placebo Comparator): RP101 matching placebo, ophthalmic sterile solution, one drop each eye every 12 h (b.i.d.) for 90 consecutive days
  Interventions: Drug: RP101

INTERVENTIONS:
Drug: RP101 — 17β-oestradiol-3-phosphate ophthalmic sterile solution
  Other Names: 17β-oestradiol-3-phosphate

SUMMARY:
The main purpose of this study is to establish whether RP101 can reduce symptoms of dry eye syndrome in post-menopausal women.

DETAILED DESCRIPTION:
Redwood Pharma is developing the novel ophthalmic product RP101 containing the known active substance 17β-oestradiol-3-phosphate and based upon the drug delivery platform IntelliGel which controls the active substance release. The novel formulation is planned to meet the still unmet medical need of an efficacious treatment against chronic dry eye in postmenopausal women.

The efficacy of the novel formulation RP101 will be investigated for the first time in the present multicentre, randomised, double-masked, parallel-group, placebo-controlled Phase II study in women post-menopausal for at least 3 years presenting with symptoms specific for dry eye syndrome of moderate to severe intensity.

The planned study will be conducted in Austria, Germany and Hungary. The primary objective of the study is to establish the effective dose/dose regimen of RP101 in these patients applying RP101 ophthalmic sterile solution or matching placebo (vehicle) once (q.d.) or twice a day (b.i.d.) for 3 months. One hundred (100) patients will be enrolled in this study. The subjects will be randomly assigned (1:1:1:1) to a treatment group and will receive one of the treatments for 90 consecutive days.

Evaluation of the clinical efficacy during and at the end of the treatment will be done on the basis of the Schirmer's test type II (with anaesthesia).

The secondary objectives of the study are:

* to evaluate the safety and tolerability of the treatment
* to evaluate the pharmacokinetics (PK) of serum 17β-oestradiol after the 1st and the last dose (only PK substudy).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: signed written informed consent before inclusion in the study
* Sex and menopause: postmenopausal women; postmenopausal condition defined as final menstrual period at least 3 years before the screening
* Dry eye syndrome: patients with moderate to severe dry eye syndrome
* Tear film breakup time: TFBUT ≤ 10 sec in the worse eye (study eye)
* Visual acuity: corrected visual acuity ≥ 20/200 in each eye
* Symptoms: at least 2 of the typical dry eye syndrome symptoms since at least 3 months before the screening: foreign body sensation, burning/stinging, redness, tearing, pain, itching, blurred vision, photophobia, eyelid swelling, moisture and mucous discharge
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study

Exclusion Criteria:

* Meibomian gland dysfunction: severe Meibomian gland dysfunction defined as lid deformity, marked lid margin hyperaemia or severe Meibomian gland loss
* Ophthalmic treatment: current use of topical ophthalmic medications other than ocular lubricants or artificial tears within 30 days before the screening
* Ocular infection and inflammation: presence of any bacterial or viral or fungal infection in either eye or active inflammation not related to dry eye disease (i.e. follicular conjunctivitis, iris or preauricular adenopathy) in either eye
* Ophthalmic diseases: severe forms of ophthalmic surface diseases e.g. ocular pemphigoid, Sjögren's disease, exposure keratitis
* Ophthalmic surgery: history of ophthalmic surgery or trauma in the last 6 months; history of laser-assisted in situ keratomileusis (LASIK) in the previous 12 months
* Diseases: uncontrolled systemic diseases including cardiovascular, pulmonary and/or renal diseases, diabetes, hypertension; history of ovarian, breast or uterine cancer or unexplained vaginal bleeding
* Investigative drug studies: participation in the evaluation of any investigational product or medical device for 30 days before this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Schirmer's test type II (with anaesthesia) | From Screening up to 90 days
  Schirmer's test uses sterile strips inserted into the eye to measure the basal aqueous tear secretion.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) for ocular tolerability (foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision, redness, tearing, eyelid swelling and photophobia) | From Screening up to 90 days
  It will be assigned by the patients using a 100 mm VAS.
Symptom assessment in Dry Eye (SANDE) | From Screening up to 90 days
  The patient symptoms of ocular dryness and/or irritation will be quantified on a Visual Analogue Scale (VAS) 0-100 mm based on two questions that inquire about both severity and frequency of symptoms. The patients will evaluate their symptoms on the VAS scale giving the value they are feeling from none (0 mm) to an extreme value (100 mm).
Visual acuity assessment using an Early Treatment Diabetic Retinopathy Study [ETDRS] chart | From Screening up to 90 days
  Best correction will be determined by careful refraction using a retroilluminated ETDRS 4 meter distance acuity chart. The correct number of letters read by the patient is recorded and evaluated.
Slit lamp examination (SLE) | From Screening up to 90 days
  The SLE will be performed before the instillation of any dilating or anaesthetic eye drops or the fluorescein agent.
TFBUT | From Screening up to 90 days
  Tear film break up time (TFBUT) will be measured by determining the time to tear break-up after instillation of sodium fluorescein solution into the inferior conjunctival culde-sac of each eye.
Fundus ophthalmoscopy | From Screening up to 90 days
  The fundus examination will include ophthalmoscopic assessments of vitreous, macula, retina and optic nerve head for both eyes.
Corneal fluorescein staining | From Screening up to 90 days
  The corneal fluorescein staining evaluates cornea and conjunctiva epithelium damage.
Treatment-emergent Adverse Event (TEAEs) | From Screening up to 104 days
  All adverse events (AEs) derived by spontaneous, unsolicited reports of the subjects, by observation and by routine open questioning will be collected and reported.
17-β-oestradiol serum concentrations | Day 1 and Day 90
  Using a fully validated analytical method.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Björklund, MSc Pharm, Study Director — Redwood Pharma AB
Locations (8):
- Medical University of Vienna - Department of Clinical Pharmacology, Vienna, Austria
- Germany (3):
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Augenheilkunde, Greifswald
  - Universitätsmedizin Mainz Augenklinik und Poliklinik Klinisches, Mainz
  - Klinikum rechts der Isar der Technischen Universität München, Anstalt des öffentlichen Rechts Klinik und Poliklinik für Augenheilkunde, München
- Hungary (4):
  - Óbudai Egészség Centrum, Budapest
  - Swan Med Hungary Kft., Létavértes
  - MacroKlinika, Miskolc
  - Mentaház Magánorvosi Központ, Székesfehérvár

REFERENCES:
- [Derived] Schmidl D, Szalai L, Kiss OG, Schmetterer L, Garhofer G. A Phase II, Multicenter, Randomized, Placebo-Controlled, Double-Masked Trial of a Topical Estradiol Ophthalmic Formulation in Postmenopausal Women with Moderate-to-Severe Dry Eye Disease. Adv Ther. 2021 Apr;38(4):1975-1986. doi: 10.1007/s12325-021-01680-3. Epub 2021 Mar 12. PMID 33710587